CLINICAL TRIAL: NCT05882071
Title: SGLT2i Use in France Based on SNDS Data Claim
Brief Title: Non-interventional Study (NIS) on Sodium-glucose Co-transporter-2 Inhibitors (SGLT2i) Use in France
Status: Active, not recruiting | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1245-0287
Record Dates: First submitted 2023-05-22; First posted 2023-05-31 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sodium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients initiating treatment with SGLT2i
  Interventions: Drug: Sodium/glucose cotransporter-2 inhibitors (SGLT2i)
- Type 2 diabetes mellitus patients initiating SGLT2i
  Interventions: Drug: Sodium/glucose cotransporter-2 inhibitors (SGLT2i)

INTERVENTIONS:
Drug: Sodium/glucose cotransporter-2 inhibitors (SGLT2i) — Sodium/glucose cotransporter-2 inhibitors (SGLT2i)

SUMMARY:
The primary objective of this study are:

- Describe the characteristics of all patients initiating sodium-glucose co-transporter-2 inhibitors (SGLT2i) and the modalities of prescriptions of these two drugs and the concomitant treatments.

The secondary objectives are:

* Assess the occurrence of atheromatous cardiovascular events (unstable angina, fatal and non-fatal Myocardial infarction (MI), Transient ischemic attack (TIA), fatal and non-fatal stroke), deaths from all causes, hospitalization for heart failure and hospitalization for end-stage renal disease as main and related diagnoses during the exposure to the studied treatment
* Assess the occurrence of the main safety events (ketoacidosis, lower limb amputation and Fournier's gangrene) during the exposure to the studied treatment

ELIGIBILITY:
Inclusion Criteria:

* population includes all patients initiating a treatment with SGLT2i between April 1, 2020, and December 31, 2024.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in France initiating a treatment with SGLT2i between April 1, 2020, and December 31, 2024.
Sampling Method: Non-Probability Sample
Enrollment: 547150 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Baseline characteristic: Age | up to 5 years
Baseline characteristic: Gender | up to 5 years
Baseline characteristic: Region of residence | up to 5 years
Baseline characteristic: History of diabetes (date of first Long Term Disease (LTD) status related to diabetes) | up to 5 years
Baseline characteristic: Type of diabetes | up to 5 years
Proportion of patients with a history of cardio-vascular events including heart failure hospitalizations and lower limb amputation, renal events, ketoacidosis, Fournier's gangrene over the two years before the index date (initiation of SGLT2i) | up to 5 years

SECONDARY OUTCOMES:
Incidence rate of acute cardiovascular atheromatous events during the exposure period following initiation of the SGLT2i | up to 5 years
Time from drug initiation to first event of acute cardiovascular atheromatous events | up to 5 years
Incidence rate of heart failure hospitalization during the exposure period following initiation of the SGLT2i | up to 5 years
Time from drug initiation to first event of heart failure hospitalization | up to 5 years
Incidence rate of deaths all cause during the exposure period following initiation of the SGLT2i | up to 5 years
Time from drug initiation to death all cause | up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Boehringer Ingelheim, Paris, France

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com